CLINICAL TRIAL: NCT07361393
Title: Application of Blood Flow Restriction Training in Cardiac Patients: CARDresfluj Study
Acronym: CARDresfluj
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Ivan Chulvi Medrano, Associate Professor of Physical Education and Sport, University of Valencia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2024-FIS-3751550
Record Dates: First submitted 2026-01-13; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Rehabilitation
Keywords: blood flow restriction
MeSH Terms: interventions — Blood Flow Restriction Therapy; Clinical Trials, Phase III as Topic; Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Flow Restriction (Experimental): A pneumatic compression cuff, calibrated to 40% of the total arterial occlusion pressure-preliminarily determined via Doppler ultrasound-will be positioned at the axillary region for the performance of biceps curls and at the inguinal region for the leg press. The training protocol will follow the established consensus of one set of 30 repetitions followed by three sets of 15 repetitions, with 60-second inter-set rest intervals during which the cuff will be deflated to allow for reperfusion
  Interventions: Other: Blood Flow Restriction Exercise
- Traditional Cardiac Rehabilitation, phase III (Active Comparator): The control group will undergo the identical intervention protocol, but without the application of blood flow restriction
  Interventions: Other: Traditional Cardiac Rehabilitation, phase III

INTERVENTIONS:
Other: Blood Flow Restriction Exercise — A pneumatic compression cuff, calibrated to 40% of the total arterial occlusion pressure-preliminarily determined via Doppler ultrasound-will be positioned at the axillary region for the performance of biceps curls and at the inguinal region for the leg press. The training protocol will follow the established consensus of one set of 30 repetitions followed by three sets of 15 repetitions, with 60-second inter-set rest intervals during which the cuff will be deflated to allow for reperfusion
  Other Names: Occlusive training
  Arms: Blood Flow Restriction
Other: Traditional Cardiac Rehabilitation, phase III — The control group will undergo the identical intervention protocol, but without the application of blood flow restriction
  Other Names: Cardiovascular Rehabilitation
  Arms: Traditional Cardiac Rehabilitation, phase III

SUMMARY:
1. Research Objective

   To describe and compare the effects on cardiovascular health, physical fitness, quality of life, oxidative stress, and sleep quality resulting from a conventional resistance training program versus a conventional resistance training program partially implemented with Blood Flow Restriction (BFR) in patients with Phase III cardiac disease.
2. Methodology, Expected Collaboration, and Duration

Participants will be invited to undergo assessments for physical fitness, functional capacity, cardiological, hemodynamic, and biochemical control, as well as perceived quality of life and sleep quality, both prior to and following the intervention.

Your collaboration in this study will consist of participating in a Phase III Cardiac Rehabilitation program, monitored by specialized personnel and supervised by a cardiologist.

The intervention is based on a resistance training program supplemented with leg press and biceps curl exercises. These specific exercises will be performed using a blood flow restriction cuff.

The intervention will be conducted twice weekly over a 10-week period, followed by a 2-months washout (rest) period. Subsequently, the 10-week intervention will be repeated; however, if the first phase was completed with the use of cuffs, the second phase will be conducted without them, and vice-versa (cross-over design).

ELIGIBILITY:
Inclusion Criteria:

* All participants must be of legal age (≥18 years) and provide signed informed consent prior to any study procedures
* Participants must have a confirmed medical diagnosis of stable cardiac disease (e.g., post-myocardial infarction, stable angina, or post-revascularization) as documented by a specialist.
* All subjects must be currently enrolled in or actively participating in a Phase III Cardiac Rehabilitation program (the maintenance phase).
* Evidence of clinical stability is required, ensuring that participants can safely perform resistance training without immediate cardiovascular contraindications.

Exclusion Criteria:

* Unstable Cardiovascular Status: Presence of unstable angina, uncontrolled cardiac arrhythmias, or severe symptomatic aortic stenosis.
* Recent Acute Events: Myocardial infarction, coronary artery bypass graft (CABG), or other major cardiac surgeries within the last 3 months (or outside the timeframe defined for Phase III eligibility).
* Uncontrolled Hypertension: Resting systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg despite pharmacological treatment.
* Specific Contraindications to BFR: History of deep vein thrombosis (DVT), peripheral vascular disease, or severe lymphedema in the limbs designated for cuff application.
* Musculoskeletal Limitations: Any orthopedic or neuromuscular condition that prevents the safe performance of biceps curls or leg press exercises.
* Concurrent High-Intensity Training: Participation in any other structured vigorous-intensity exercise program that could confound the results of the intervention.
* Medical Instability: Significant comorbid conditions, such as uncontrolled metabolic disease (e.g., Type 2 Diabetes with severe complications), advanced renal failure, or respiratory diseases that limit functional capacity below the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Indirect 1 repetition maximum | Pre intervention (week 0) and post intervention (week 11) in experimental and control phases
  The Brzycki formula is a widely recognized equation used to predict a participant's maximum strength based on submaximal performance. Similar to the Epley method, it is highly valued in clinical settings-such as Phase III Cardiac Rehabilitation-because it avoids the excessive cardiovascular strain and the Valsalva maneuver associated with maximal (1RM) testing.
  Procedure and ProtocolSubmaximal Loading: A load is selected that the participant can lift for a range of 2 to 10 repetitions. Research suggests that the Brzycki formula maintains higher accuracy when the number of repetitions is kept below 10.
  1Execution to Volitional Fatigue: The participant performs the exercise (e.g., leg press or biceps curl) with controlled technique until they reach a point where no further complete repetitions can be performed.
  Calculation: The achieved repetitions and the weight used are integrated into the formula to determine the theoretical 1RM.
Heart Rate Variability | Pre intervention (week 0) and post intervention (week 11) in experimental and control phases
  Heart Rate Variability (HRV) will be monitored to evaluate the balance between sympathetic and parasympathetic nervous system activity. The Polar H10 heart rate monitor-a chest-strap based sensor-will be utilized to capture R-R intervals (the time between successive heartbeats) with high temporal resolution.
  Data Acquisition Protocol Preparation: To ensure optimal conductivity and signal quality, the electrode areas of the Polar H10 strap will be moistened with water or conductive gel before being secured firmly around the participant's chest, just below the pectoral muscles.
  Stabilization Period: Participants will remain in a seated position for a 15-minute stabilization period to achieve a resting physiological state and minimize external artifacts.
  Recording: R-R interval data will be recorded for a duration of whole session and 15 minutes post-session
  Signal Processing: The raw data will be filtered using a compatible software interface (e.g., Kubios HRV).
Tendon Thickness | Pre intervention (week 0) and post intervention (week 11) in experimental and control phases
  To evaluate structural adaptations following the intervention, the tendon thickness of the biceps brachii and the quadriceps femoris (specifically the patellar tendon) was measured using high-resolution B-mode ultrasonography. This non-invasive imaging technique allows for the precise quantification of connective tissue morphology.
  Measurement ProtocolBiceps Brachii Tendon: Measurements were taken with the participant in a supine position, with the arm fully extended and supinated. The transducer was placed longitudinally over the bicipital groove of the humerus to identify the long head of the biceps tendon.
  Quadriceps Femoris (Patellar Tendon): The participant was placed in a supine position with the knee flexed at 30% to maintain tendon tension and eliminate slack. The measurement was localized at proximal region of the patella.
  Data Acquisition: Images were captured in the longitudinal and transversal plane.

SECONDARY OUTCOMES:
CSA grossor | Pre intervention (week 0) and post intervention (week 11) in experimental and control phases
  Muscle Thickness and Cross-Sectional Area (CSA) were measured using high-resolution B-mode ultrasonography. Specifically, the biceps brachii and the rectus femoris were assessed at standardized anatomical landmarks.
  Measurement Sites and Protocol for Biceps Brachii: Measurements were taken at two-thirds of the distance from the acromion process to the cubital fossa (lateral epicondyle). This site ensures the measurement captures the muscle at its maximum morphological development.
  Rectus Femoris: The assessment was conducted at two-thirds of the distance between the anterior superior iliac spine (ASIS) and the superior border of the patella. This distal measurement site is highly sensitive to changes in muscle architecture during resistance training.
  Technique: The ultrasound transducer was placed perpendicular to the longitudinal axis of the muscle. Minimal pressure was applied to the skin to avoid tissue compression, which could lead to an underestimation of thickness.
Blood Pressure | Pre intervention (week 0) and post intervention (week 11) in experimental and control phases
  Resting arterial blood pressure (BP)-specifically Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)-was measured using a digital oscillometric sphygmomanometer (Omron Healthcare, Inc.). This non-invasive method was utilized to monitor hemodynamic stability throughout the study duration. The blood pressure assessment followed the standardized clinical procedures detailed in the American Heart Association (AHA) guidelines for blood pressure measurement in humans. This rigorous adherence ensured the minimization of observer bias and controlled for external factors that could influence hemodynamic readings.
Handgrip test | Pre intervention (week 0) and post intervention (week 11) in experimental and control phases
  Handgrip strength (HGS) was measured using a calibrated hydraulic dynamometer (e.g., Jamar or similar) to evaluate maximal isometric upper-body strength. This test serves as a reliable proxy for total muscle strength and is a critical functional marker in Phase III Cardiac Rehabilitation. Participants were instructed to exert their maximum grip force for 3 to 5 seconds. Strong verbal encouragement was provided to ensure peak effort ("Squeeze, squeeze, squeeze!").
Timed-uo and Go | Pre intervention (week 0) and post intervention (week 11) in experimental and control phases
  Functional mobility and dynamic balance will be assessed using the Timed Up and Go (TUG) test. Following standardized clinical protocols, participants start seated in a standard armchair (approx. 46 cm high). On the "go" command, they rise, walk at a comfortable and safe pace to a line marked 3 meters away, turn, return to the chair, and sit down.
  Timing starts at the signal and stops when the participant's back touches the backrest. To ensure reliability, a practice trial will be performed, followed by two recorded trials, using the average time for analysis. This test is a validated predictor of fall risk and functional independence in Phase III cardiac patients. All procedures will be supervised to ensure participant safety, particularly during the turn and sitting phases.
30 seconds sit to stand | Pre intervention (week 0) and post intervention (week 11) in experimental and control phases
  The 30-second Sit-to-Stand test will be used to assess proximal lower-limb functional strength and endurance. Following the established protocol, the participant sits in the middle of a chair (approx. 43-45 cm high) with a flat backrest, feet shoulder-width apart, and arms crossed over the chest.
  On the "start" command, the participant rises to a full standing position and returns to a full sit as many times as possible within 30 seconds. The score is the total number of completed stands; if the participant is over halfway to a standing position when time expires, it counts as a full stand. This test is a validated clinical tool for cardiac populations, reflecting the ability to perform activities of daily living. A demonstration and a brief practice of two repetitions will precede the final assessment to ensure proper technique and safety.
6 min walking | Pre intervention (week 0) and post intervention (week 11) in experimental and control phases
  Submaximal exercise capacity will be assessed using the 6-Minute Walk Test (6MWT) in accordance with the American Thoracic Society (ATS) guidelines. The test will be performed on a flat, 30-meter indoor corridor. Participants are instructed to walk as far as possible for six minutes at their own pace, being permitted to slow down or rest if necessary. The total distance covered (6MWD) in meters will be recorded as the primary outcome. This test is highly sensitive to changes in functional status and is a gold-standard prognostic marker in Phase III cardiac rehabilitation. A technician will supervise the test with emergency equipment available to ensure patient safety.
SF-36 | Pre intervention (week 0) and post intervention (week 11) in experimental and control phases
  Health-related quality of life (HRQoL) will be assessed using the Short Form-36 (SF-36) Health Survey, a widely validated multidimensional instrument. This questionnaire consists of 36 items that evaluate eight health domains: physical functioning, physical role limitations, bodily pain, general health perceptions, vitality, social functioning, emotional role limitations, and mental health.
  Results are aggregated into two primary summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Scores for each domain range from 0 to 100, where higher scores represent superior perceived health status. The SF-36 is highly sensitive to the effects of exercise interventions in cardiac populations. Participants will complete the survey in a quiet environment to minimize external influence, ensuring the capture of reliable subjective data regarding their well-being.

OTHER OUTCOMES:
Assessment of Sleep Quality: Pittsburgh Sleep Quality Index (PSQI) | Pre intervention (week 0) and post intervention (week 11) in experimental and control phases
  Sleep quality will be evaluated using the Pittsburgh Sleep Quality Index (PSQI), a validated self-report questionnaire that assesses sleep patterns over a one-month interval. The instrument consists of 19 individual items grouped into seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
  Each component is scored from 0 to 3, yielding a global score ranging from 0 to 21. A global score greater than 5 indicates "poor" sleep quality. The PSQI is highly reliable for identifying sleep disorders in clinical populations, including those in cardiac rehabilitation. Participants will complete the questionnaire in a controlled, quiet setting to ensure accuracy. This assessment allows for the objective quantification of how the exercise intervention and blood flow restriction may influence restorative sleep.
IPAC | Pre intervention (week 0) and post intervention (week 11) in experimental and control phases
  Physical activity levels will be assessed using the International Physical Activity Questionnaire (IPAQ) - Short Form. This validated instrument quantifies the duration and frequency of walking, moderate-intensity, and vigorous-intensity activities performed during the previous seven days.
  Data will be processed following the official IPAQ scoring protocol, converting reported activities into Metabolic Equivalent of Task minutes per week (MET-min/week). Participants will be categorized into three activity levels: low, moderate, or high. The IPAQ is a standardized tool widely used in clinical research to monitor lifestyle changes. In this study, it allows for the control of external physical activity levels that might influence the cardiovascular and musculoskeletal adaptations observed during the Phase III Cardiac Rehabilitation program.

IPD SHARING:
Plan to Share IPD: Undecided